CLINICAL TRIAL: NCT04413162
Title: Measurement of Shoulder Range of Motion Using Microsoft Kinect 2.0 in Patients Undergoing Ultrasound-guided Capsular Distension for Adhesive Capsulitis
Brief Title: Using Kinect Motion Capture to Measure Shoulder Motion in Patients Undergoing Capsular Distension for Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1490166
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-11

CONDITIONS: Adhesive Capsulitis; Adhesive Capsulitis of Shoulder; Frozen Shoulder; Shoulder Frozen; Shoulder Pain; Mobility Limitation
Keywords: adhesive capsulitis; frozen shoulder; shoulder pain; range of motion; capsular distention; capsular distension
MeSH Terms: conditions — Bursitis; Shoulder Pain; Mobility Limitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- measurement before and after capsular distention (Other)
  Interventions: Other: Kinect motion tracking system

INTERVENTIONS:
Other: Kinect motion tracking system — Kinect motion tracking system is used to measure shoulder range of motion compared to goniometric measurement.

SUMMARY:
This study will compare shoulder range of motion assessment using the Kinect motion tracking system vs goniometer in patients with adhesive capsulitis (frozen shoulder) undergoing ultrasound-guided capsular distention procedures (standard of care).

The investigators hypothesize that, for shoulder adhesive capsulitis, the Kinect Motion Analysis 2.0 system will provide reliable results in a shorter and more efficient amount of time in comparison to traditional goniometer methods.

DETAILED DESCRIPTION:
The study will be a single-center, investigator-initiated protocol to assess the reliability of the Kinect Motion Analysis 2.0 Motion Tracking System for Range Of Motion (ROM) assessment in patients with Shoulder Adhesive Capsulitis undergoing ultrasound guided capsular distention procedures (standard of care for adhesive capsulitis). Secondarily, the study will describe the relationship between range of motion of the shoulder girdle in the four quadrants of normalized reachable workspace by the Kinect 2.0, PROMIS person-reported outcome scores for pain, pain interference and function (general mobility and upper extremity function), and VAS pain scores.

Study participants are anticipated to remain in the study for 12 weeks: an initial visit followed by 6- and 12-week follow up visits. Given the nature of scheduling appointments in medical clinics, 12 weeks is an approximation; the actual duration may occasionally be 1-2 weeks longer if needed to successfully complete the follow-up visit.

The investigators hypothesize that, for shoulder adhesive capsulitis, the Kinect Motion Analysis 2.0 system will provide reliable results in a shorter and more efficient amount of time in comparison to traditional goniometer methods.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of limited ROM due to adhesive capsulitis
2. duration of symptoms of ≥ 3 months
3. persistent functional limitation (defined as either limitations occupationally, in independent activities of daily living, or activities of daily living)
4. X-rays and MRI excluding alternative diagnosis
5. age 18 years or older.

Exclusion Criteria:

1. prior shoulder surgery on the affected side
2. complete rotator cuff tear (based on clinical history, examination, and imaging) or planned surgical intervention on the affected side
3. ipsilateral subacromial injection within the last 3 months
4. autoimmune or rheumatologic disease affecting the joints
5. lack of scheduled same-day physical therapy appointment
6. inability to complete follow-up appointments or surveys
7. inability to provide informed consent
8. symptomatic glenohumeral or acromioclavicular pathology
9. referred pain from the neck or internal organs
10. generalized myofascial pain syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
change in shoulder range of motion | 12 weeks
  measured in degrees (high number of degrees = better range of motion)

SECONDARY OUTCOMES:
PROMIS score - upper extremity | 12 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) is a validated, 46-item, self-reported system to assess physical function and symptoms in patients with disorders of the limb. Range of possible values: 46-230. (Higher score indicates higher function and outcomes)
DASH score | 12 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 38-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities. Range of possible values: 38-150. (Lower score indicates better function / less disability)
VAS score | 12 weeks
  Visual analog scale is a validated, subjective measure for pain. Range of possible values: 0-10. (Higher score indicates more pain)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Mullins, MD, Principal Investigator — UC Davis Health
Locations (1):
- UC Davis Sports Medicine, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/using-kinect-motion-capture-to-measure-shoulder-motion-for-capsular-distension-in-adhesive-capsulitis-frozen-shoulder-654329/